CLINICAL TRIAL: NCT05620108
Title: Intubating Conditions at Various Levels of Neuromuscular Blockade
Brief Title: Intubating Conditions of Neuromuscular Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-009153
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intubation at TOFC=1 (Experimental): Subjects scheduled for an elective surgical procedure will have endotracheal intubation performed when muscles are almost relaxed and monitoring shows only a single count of muscle twitch (in response to a monitor that assesses muscle relaxation)
  Interventions: Procedure: Endotracheal Intubation at TOFC=1
- Intubation 2 minutes after rocuronium administration (Active Comparator): Subjects scheduled for an elective surgical procedure will have endotracheal intubation performed 2 minutes after the anesthesia provider gives muscle relaxing medication
  Interventions: Procedure: Endotracheal Intubation 2 minutes after rocuronium administration

INTERVENTIONS:
Procedure: Endotracheal Intubation at TOFC=1 — Intubation using a video laryngoscopy will be performed after train-of-four (TOFC) stimulation indicates neuromuscular blockade
  Arms: Intubation at TOFC=1
Procedure: Endotracheal Intubation 2 minutes after rocuronium administration — Intubation using a video laryngoscopy will be performed 2 minutes after administration of rocuronium at 0.6 mg/kg (usual current clinical routine)
  Arms: Intubation 2 minutes after rocuronium administration

SUMMARY:
The purpose of this research is to learn about the difference in the endotracheal intubation condition (ease of using a device to view vocal cords, position of vocal cords, and patient's reaction to endotracheal tube insertion) and determining the appropriate time to perform the intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate and provide an informed consent.
* Patients undergoing elective surgical procedures that require use of NMBA agents (rocuronium) administered intraoperatively.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis.
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents; i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm into the sterile field.
* Patients receiving a rapid sequence induction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Intubation at TOFC=1: Subjects scheduled for an elective surgical procedure had endotracheal intubation performed when muscles were almost relaxed and monitoring showed only a single count of muscle twitch (in response to a monitor that assessed muscle relaxation)
  Endotracheal Intubation at TOFC=1: Intubation using a video laryngoscopy was performed after train-of-four (TOFC) stimulation indicated neuromuscular blockade
- Intubation 2 Minutes After Rocuronium Administration: Subjects scheduled for an elective surgical procedure had endotracheal intubation performed 2 minutes after the anesthesia provider gave muscle relaxing medication
  Endotracheal Intubation 2 minutes after rocuronium administration: Intubation using a video laryngoscopy was performed 2 minutes after administration of rocuronium at 0.6 mg/kg (usual current clinical routine)
Period: Overall Study
Arm/Group | Intubation at TOFC=1 | Intubation 2 Minutes After Rocuronium Administration
Started | 85 | 85
Completed | 84 | 83
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubation at TOFC=1 | Intubation 2 Minutes After Rocuronium Administration | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (12.9) | 59.1 (14.8) | 59.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 45 | 47 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 80 | 78 | 158
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 79 | 78 | 157
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Optimal Intubating Conditions
Description: The number of subjects who had optimal intubating conditions (total composite score of 3) will be evaluated by the healthcare providers using a scale that includes 3 variables (ease of laryngoscopy, vocal cord position, and reaction to tracheal tube insertion) with 3 response options per each evaluation. The composite score (1-3) will be used, with the lowest total score of 3 correlating with optimal intubating conditions and the highest score of 9 representing the worse possible intubating conditions.
Time Frame: Approximately 15 minutes after intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Intubation at TOFC=1 | Intubation 2 Minutes After Rocuronium Administration
Number analyzed (Participants) | 84 | 83
Participants | 61 | 47
Statistical Analysis 1: Comparison: Intubation at TOFC=1 vs Intubation 2 Minutes After Rocuronium Administration; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 15 minutes.
Description: Adverse events were collected through specific questioning and examination.
Arm/Group | Intubation at TOFC=1 | Intubation 2 Minutes After Rocuronium Administration
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05620108/Prot_SAP_000.pdf